CLINICAL TRIAL: NCT02421003
Title: Exploratory Study, Prospective, of Volume, Composition and Bacteriology of the Recovered Blood of Multi-perforated Catheter Inserted in the Drapes Thickness of Incisional Sternal Area During Heart Surgery
Acronym: Blood-in-drape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2014_843_0017
Record Dates: First submitted 2015-04-10; First posted 2015-04-20 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Heart Surgery
Keywords: heart surgery blood
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Patients undergoing heart surgery
  Interventions: Procedure: heart surgery

INTERVENTIONS:
Procedure: heart surgery

SUMMARY:
The recovered blood into the surgical site at the border of the fields, is very rich in red blood cells, due to the adjacency of the bone marrow and the sternum.

The blood recovered from the surgical site at the border of the fields, is richer in red blood cells than the bloodstream of the patient.

The recovered blood into the surgical site at the border of the fields, is not contaminated and bacteriological cultures are negative.

Consequences: The recovered blood in the surgical site at the edge of fields, can be recovered in the Saver® Cell for reprocessing and re-injected into the patient.

There isn't in our knowledge of published clinical data on the volume and composition of the recovered blood in the surgical site after cardiac surgery.

The analysis of the available literature does not allow to estimate the expected outcomes us. Therefore, this study will be exploratory in nature and will aim to estimate the volume and the content of red blood cells from blood recovered, and generate clinical data to be used in subsequent confirmatory tests.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Any open heart surgery with or without extracorporeal circulation
* Signature of informed consent
* Affiliation to social security

Exclusion Criteria:

* Subjects legally protected or unable to consent
* Persons deprived of liberty
* Cardiac Surgery extreme emergency (due to difficulties obtaining informed consent)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measurement of red blood cell numeration from blood collected. | Between the incision and the closure.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles TOUATI, Doctor, Principal Investigator — CHU Amiens
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France